CLINICAL TRIAL: NCT02950636
Title: Effect of Yoga on Mood and Quality of Life in Patients With Refractory Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140045; UL1TR000001 (NIH)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Depression; Anxiety
Keywords: Epilepsy
MeSH Terms: conditions — Depression; Anxiety Disorders; Epilepsy | interventions — Yoga

ARMS (1):
- Restorative Yoga (Experimental): Subjects will participate in a structured restorative yoga program. Subjects will attend a 60 minute restorative yoga class twice a week for 8 weeks in a yoga studio.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Restorative Yoga

SUMMARY:
The purpose of this study is to learn if a structured yoga program can reduce anxiety, improve depression, and improve quality of life in patients with medication resistant epilepsy (MRE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral or bilateral temporal lobe epilepsy
* Presence 3 or more seizures per month
* No medical contraindications to yoga
* Willing and able to perform simple non strenuous yoga exercises
* Ability to get on the floor and up again without assistance
* Ambulatory
* Ability to travel to the yoga class twice a week

Exclusion Criteria:

* Any yoga in the last 6 months
* Inability to perform yoga exercises
* History of epilepsy surgery within the last year
* Currently pregnant or less than 6 week postpartum

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) | Change from Week 4 to Week 12
  The NDDI-E is a 6 item questionnaire. Scores for each question range from 1 (never) to 4 (all the time). There is a maximum score of 24. The higher the score the more severe the depression.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7-item (GAD-7) scale | Change from Week 4 to Week 12
  The GAD-7 is a 7 item questionnaire. Scores for each question range from 0 (not at all) to 3 (nearly every day). There is a maximum score of 21. The higher the score the more severe the anxiety. A score over 15 represents severe anxiety. A score under 10 may indicate GAD and would prompt further examination.
Change in Quality of Life in Epilepsy-Patient-Weighted (QOLIE-31-p) | Change from Baseline to Week 12
  The QOLIE-31-p is a 38 item questionnaire. Scores range from 0-100. Higher scores relate to higher distress.
Frequency of seizures | Week 12
  Count of seizures in study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Hammond, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States